CLINICAL TRIAL: NCT04917861
Title: A Phase 2, Randomized, Observer-Blind, Placebo-Controlled, Dose Confirmation Study to Evaluate the Safety, Tolerability, and Immunogenicity of Zika Vaccine mRNA-1893 in Adults Aged 18 Through 65 Years and Living in Endemic and Non-Endemic Flavivirus Areas
Brief Title: A Study of Zika Vaccine mRNA-1893 in Adult Participants Living in Endemic and Non-Endemic Flavivirus Areas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1893-P201; HHSO100201600029C (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Zika Virus
Keywords: Flavivirus; mRNA-1893; Zika vaccine; Moderna
MeSH Terms: conditions — Zika Virus Infection | interventions — GLS-5700 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mRNA-1893 Low Dose (2-Dose Regimen) (Experimental): Participants will receive mRNA-1893 at a low dose level administered as a 2-dose regimen with 28-day (-3/+7 days) interval between vaccinations (administered on Day 1 and Day 29).
  Interventions: Biological: mRNA-1893
- mRNA-1893 High Dose (2-Dose Regimen) (Experimental): Participants will receive mRNA-1893 at a high dose level administered as a 2-dose regimen with 28-day (-3/+7 days) interval between vaccinations (administered on Day 1 and Day 29).
  Interventions: Biological: mRNA-1893
- mRNA-1893 High Dose (1-Dose Regimen) (Experimental): Participants will receive placebo matching to mRNA-1893 on Day 1 and mRNA-1893 at a high dose level administered as a 1-dose regimen (administered on Day 29). There will be 28-day (-3/+7 days) interval between vaccinations.
  Interventions: Biological: mRNA-1893; Biological: Placebo
- Placebo (Placebo Comparator): Participants will receive placebo matching to mRNA-1893 administered as a 2-dose regimen with 28-day (-3/+7 days) interval between vaccinations (administered on Day 1 and Day 29).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1893 — Solution for injection
  Other Names: Zika vaccine
  Arms: mRNA-1893 High Dose (1-Dose Regimen); mRNA-1893 High Dose (2-Dose Regimen); mRNA-1893 Low Dose (2-Dose Regimen)
Biological: Placebo — 0.9% sodium chloride solution for injection
  Arms: Placebo; mRNA-1893 High Dose (1-Dose Regimen)

SUMMARY:
This clinical study will evaluate the safety, tolerability, and reactogenicity of 2 dose levels of messenger RNA (mRNA)-1893 Zika vaccine in comparison to a placebo control in healthy participants who are flavivirus-seronegative and in participants who are flavivirus-seropositive.

ELIGIBILITY:
Key Inclusion Criteria:

* Understands and agrees to comply with the study procedures and provides written informed consent.
* According to investigator assessment, is in good general health and can comply with study procedures.
* Female participants of childbearing potential may be enrolled in the study if the participant: has a negative pregnancy test at the Eligibility Visit and on the day of the first investigational product (IP) injection; has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first IP injection; has agreed to continue adequate contraception through 3 months following the last IP injection; and is not currently breastfeeding.

Key Exclusion Criteria:

* Participant is acutely ill or febrile (temperature ≥38.0°Celsius/100.4°Farenheight) on the day of the first or second vaccination.
* Participant had prior administration of a ZIKV vaccine candidate during a clinical study investigation.
* Participant had prior administration of a marketed dengue vaccine or dengue vaccine candidate under clinical study investigation.
* Participant has a body mass index (BMI) from ≤18 or ≥35 kilograms (kg)/square meter (m^2).
* Participant has a history of myocarditis, pericarditis, or myopericarditis.
* Participant has a history of a diagnosis or condition that, in the judgement of the investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures. "Clinically unstable" is defined as a diagnosis or condition requiring significant changes in management or medication within the 2 months prior to screening and includes ongoing work-up of an undiagnosed illness that could lead to a new diagnosis or condition.
* Participant has any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that in the opinion of the investigator, might pose a risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has as a history of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine, including an mRNA vaccine or any components of an mRNA vaccine.
* Participant has received or plans to receive a nonstudy vaccine (including authorized or approved vaccines for the prevention of COVID-19) ≤28 days prior to the first IP injection or within 28 days prior to or after any IP injection. Licensed influenza vaccine received within 14 days prior to the first IP injection or plans to receive a licensed influenza vaccine 14 days prior to through 14 days following each IP injection are not exclusionary.
* Participant has received systemic immunoglobulins or blood products within 3 months prior to the day of enrollment.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days of the Day 1 Visit.
* Participant has participated in an interventional clinical study within 28 days prior to the day of enrollment or plans to do so while enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - Meridian Clinical Research (Sioux City, IA), Sioux City, Iowa
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Benchmark Research - Fort Worth, Fort Worth, Texas
- Puerto Rico (7):
  - Clinical Research Puerto Rico, Inc., Guayama, PR
  - Ponce Medical School Foundation, Inc., Ponce, PR
  - Clinical Research Puerto Rico, Inc., San Juan, PR
  - Latin Clinical Trial Center, Inc., San Juan, PR
  - GCM Medical Group, PSC, San Juan, PR
  - Carribean Medical Research, San Juan, PR
  - University of Puerto Rico, San Juan, PR

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 808 participants were enrolled. One participant was randomized at two sites and received two injections. This participant was not presented under Per-Protocol Set but kept in Full Analysis Set, Safety Set, and Solicited Safety Set. This participant was discontinued from the study at one site upon the discovery of the duplicate participation and the incident was documented.
Groups:
- Placebo: Participants received placebo matched to mRNA-1893 administered as a 2-dose regimen with 28-day interval between vaccinations (administered on Day 1 and Day 29).
- mRNA-1893 Low Dose (2-Dose Regimen): Participants received mRNA-1893 at a low dose level administered as a 2-dose regimen with 28-day interval between vaccinations (administered on Day 1 and Day 29).
- mRNA-1893 High Dose (2-Dose Regimen): Participants received mRNA-1893 at a high dose level administered as a 2-dose regimen with 28-day interval between vaccinations (administered on Day 1 and Day 29).
- mRNA-1893 High Dose (1-Dose Regimen): Participants received placebo matched to mRNA-1893 on Day 1 and mRNA-1893 at a high dose level administered as a 1-dose regimen (administered on Day 29). There was 28-day interval between vaccinations.
Period: Main Study (196 Days)
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Started | 203 | 201 | 203 | 201
Received First Injection | 201 | 201 | 202 | 198
Received Second Injection | 187 | 188 | 187 | 191
Randomized at Second Site (Randomized to mRNA-1893 High Dose (2-Dose Regimen) and then mRNA-1893 Low Dose (2-Dose Regimen)) | 0 | 1 | 0 | 0
Completed | 173 | 166 | 176 | 178
Not Completed | 30 | 35 | 27 | 23
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 14 | 26 | 20 | 11
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 7 | 6 | 8
Not completed — Other Than Specified | 1 | 0 | 1 | 2
Period: Extension Period (Day 197 to Day 700)
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Started | 113 | 109 | 104 | 116
Completed | 97 | 96 | 89 | 93
Not Completed | 16 | 13 | 15 | 23
Not completed — Lost to Follow-up | 8 | 3 | 5 | 11
Not completed — Pregnancy | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 8 | 8 | 10
Not completed — Other Than Specified | 1 | 0 | 1 | 1
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who were randomized and received any study injection. One participant who was randomized at two sites and received two injections, has been included only once here for reporting the 'Baseline Characteristics' data. This participant was kept in both arms (Randomized to mRNA-1893 High Dose [2-Dose Regimen] and mRNA-1893 Low Dose [2-Dose Regimen]) in Full Analysis Set, Safety Set, and Solicited Safety Set for collection and reporting data.
Groups:
- mRNA-1893 High Dose (1-Dose Regimen) (: Participants received placebo matched to mRNA-1893 on Day 1 and mRNA-1893 at a high dose level administered as a 1-dose regimen (administered on Day 29). There was 28-day interval between vaccinations.
- Total: Total of all reporting groups
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen) ( | Total
Number analyzed (Participants) | 201 | 201 | 202 | 198 | 802
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 201 | 201 | 202 | 198 | 802
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 119 | 119 | 114 | 463
  Male | 90 | 82 | 83 | 84 | 339
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 106 | 106 | 110 | 107 | 429
  Not Hispanic or Latino | 94 | 94 | 91 | 90 | 369
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 167 | 167 | 174 | 172 | 680
  Race: Black or African American | 28 | 25 | 22 | 21 | 96
  Race: Asian | 0 | 2 | 1 | 2 | 5
  Race: American Indian or Alaska Native | 0 | 3 | 2 | 2 | 7
  Race: Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Race: Multiracial | 3 | 1 | 2 | 1 | 7
  Race: Other | 1 | 3 | 1 | 0 | 5
  Race: Not reported | 1 | 0 | 0 | 0 | 1
Seroresponse [Count of Participants; unit: Participants]
  Flavivirus Seronegative Participants | 96 | 92 | 105 | 111 | 404
  Flavivirus Seropositive Participants | 102 | 103 | 94 | 82 | 381
  Missing | 3 | 6 | 3 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were collected in the electronic diary. Local ARs included: pain, erythema (redness), swelling/induration (hardness). Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, body temperature (potentially fever), and chills. A summary of all serious adverse events (SAEs) and all nonserious adverse events (AEs) ("Other"), regardless of causality, is in Reported "Adverse Events" section.
Time Frame: Up to 7 days post-vaccination
Population: The Solicited Safety Set included all participants who were randomized, received any study injection, and contributed with any solicited AR data. One participant who was randomized at two sites and received two injections was kept in both arms (Randomized to mRNA-1893 High Dose [2-Dose Regimen] and mRNA-1893 Low Dose [2-Dose Regimen]) in Solicited Safety Set for collection and reporting data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 200 | 201 | 201 | 198
Participants | 86 | 164 | 183 | 163

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Unsolicited AEs were AEs that were not included in the protocol-defined solicited ARs. A treatment-emergent adverse event (TEAE) was defined as any AE not present before exposure to vaccine or any AE already present that worsened in intensity or frequency after exposure. A summary of all SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to 28 days post-vaccination
Population: The Safety Set included all participants who were randomized and received any study injection. One participant who was randomized at two sites and received two injections was kept in both arms (Randomized to mRNA-1893 High Dose [2-Dose Regimen] and mRNA-1893 Low Dose [2-Dose Regimen]) in Safety Set for collection and reporting data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 201 | 202 | 202 | 198
Participants | 39 | 47 | 52 | 45

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), AEs of Special Interest (AESIs)
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, was a congenital anomaly/birth defect, or was an important medical event. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor were required. A summary of all SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Day 1 through Day 196 for Main Study and Day 197 through Day 700 for Extension Period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Main Study: Placebo: Participants received placebo matched to mRNA-1893 administered as a 2-dose regimen with 28-day interval between vaccinations (administered on Day 1 and Day 29).
- Main Study: mRNA-1893 Low Dose (2-Dose Regimen): Participants received mRNA-1893 at a low dose level administered as a 2-dose regimen with 28-day interval between vaccinations (administered on Day 1 and Day 29).
- Main Study: mRNA-1893 High Dose (2-Dose Regimen): Participants received mRNA-1893 at a high dose level administered as a 2-dose regimen with 28-day interval between vaccinations (administered on Day 1 and Day 29).
- Main Study: mRNA-1893 High Dose (1-Dose Regimen): Participants received placebo matched to mRNA-1893 on Day 1 and mRNA-1893 at a high dose level administered as a 1-dose regimen (administered on Day 29). There was 28-day interval between vaccinations.
- Extension Period: Placebo; Extension Period: mRNA-1893 Low Dose (2-Dose Regimen); Extension Period: mRNA-1893 High Dose (2-Dose Regimen); Extension Period: mRNA-1893 High Dose (1-Dose Regimen): Participants were followed up for up to Day 700 in the extension period.
Arm/Group | Main Study: Placebo | Main Study: mRNA-1893 Low Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (1-Dose Regimen) | Extension Period: Placebo | Extension Period: mRNA-1893 Low Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 201 | 202 | 202 | 198 | 113 | 109 | 104 | 116
Participants
  SAEs | 5 | 2 | 4 | 7 | 5 | 4 | 5 | 7
  AESIs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Medically Attended AEs (MAAEs)
Description: An MAAE was an AE that led to an unscheduled visit to a healthcare practitioner. Note that the generation of the tables for the MAAE data for the Main Study occurred after the start of the Extension Period. Therefore, some of the MAAE data for this outcome measure may appear both in the Main Study and the Extension Period. A summary of all SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Day 1 through Day 196 for Main Study and Day 197 through Day 700 for Extension Period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Placebo | Main Study: mRNA-1893 Low Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (1-Dose Regimen) | Extension Period: Placebo | Extension Period: mRNA-1893 Low Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 201 | 202 | 202 | 198 | 113 | 109 | 104 | 116
Participants | 62 | 50 | 62 | 63 | 29 | 24 | 30 | 31

5. Primary Outcome: Geometric Mean Titer (GMT) of Zika Virus (ZIKV)-Specific Neutralizing Antibodies (nAbs) at Day 57, as Measured by 50% Plaque Reduction Neutralization Test (PRNT50)
Description: Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5 * LLOQ. Values that were greater than the upper limit of quantification (ULOQ) were converted to the ULOQ. LLOQ=91; ULOQ=24814. 95% confidence interval (CI) was calculated based on the t-distribution of the log-transformed values, then back transformed to the original scale for presentation.
Time Frame: Day 57
Population: The Per-Protocol Set for Antibody-Mediated Immunogenicity (PPAMI) included all participants who received any study injection, who did not have major protocol deviations that impacted AMI response, and who complied with the injection schedule and the timing of immunogenicity blood sampling to have post-injection results available for at least 1 assay component of AMI at the corresponding visit. Here, 'Number analyzed' = participants evaluable for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
titer
  All Participants | 61.06 [54.07 to 68.96] | 427.53 [343.28 to 532.45] | 434.92 [343.63 to 550.46] | 163.28 [122.68 to 217.30]
  Flavivirus-seronegative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Flavivirus-seronegative Participants | 45.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 327.95 [246.98 to 435.47] | 363.03 [277.84 to 474.35] | 68.96 [55.94 to 85.02]
  Flavivirus-seropositive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Flavivirus-seropositive Participants | 79.46 [63.92 to 98.78] | 539.17 [385.76 to 753.59] | 502.11 [337.76 to 746.45] | 558.49 [336.21 to 927.73]
Statistical Analysis 1: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; Geometric Mean Ratio (GMR) = 7.002, 95% CI 2-sided [5.451 to 8.992] — GMR (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 2: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; GMR = 7.123, 95% CI 2-sided [5.467 to 9.279] — GMR (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 3: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; GMR = 2.674, 95% CI 2-sided [1.961 to 3.646] — GMR (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 4: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; GMR = 7.208, 95% CI 2-sided [5.428 to 9.571] — GMR (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-seronegative participants
Statistical Analysis 5: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; GMR = 7.979, 95% CI 2-sided [6.106 to 10.425] — GMR (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-seronegative participants
Statistical Analysis 6: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; GMR = 1.516, 95% CI 2-sided [1.229 to 1.869] — GMR (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-seronegative participants
Statistical Analysis 7: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; GMR = 6.785, 95% CI 2-sided [4.562 to 10.092] — GMR (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-seropositive participants
Statistical Analysis 8: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; GMR = 6.319, 95% CI 2-sided [4.030 to 9.909] — GMR (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-seropositive participants
Statistical Analysis 9: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; GMR = 7.028, 95% CI 2-sided [4.056 to 12.180] — GMR (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-seropositive participants

6. Primary Outcome: GMT of ZIKV-specific nAbs at Day 57, as Measured by 80% Plaque Reduction Neutralization Test (PRNT80)
Description: Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values that were greater than the ULOQ were converted to the ULOQ. LLOQ=91; ULOQ=24814. 95% CI was calculated based on the t-distribution of the log-transformed values, then back transformed to the original scale for presentation.
Time Frame: Day 57
Population: The PPAMI included all participants who received any study injection, who did not have major protocol deviations that impacted AMI response, and who complied with the injection schedule and the timing of immunogenicity blood sampling to have post-injection results available for at least 1 assay component of AMI at the corresponding visit. Here, 'Number analyzed' = participants evaluable for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
titer
  All Participants | 20.80 [18.60 to 23.26] | 110.52 [88.59 to 137.88] | 111.21 [88.04 to 140.48] | 48.36 [36.56 to 63.97]
  Flavivirus-seronegative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Flavivirus-seronegative Participants | 16.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 69.64 [54.81 to 88.48] | 87.45 [70.01 to 109.24] | 19.89 [17.05 to 23.21]
  Flavivirus-seropositive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Flavivirus-seropositive Participants | 25.60 [20.88 to 31.38] | 166.23 [117.69 to 234.80] | 139.57 [91.83 to 212.13] | 174.18 [104.33 to 290.79]
Statistical Analysis 1: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; GMR = 5.312, 95% CI 2-sided [4.149 to 6.802] — GMR (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 2: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; GMR = 5.346, 95% CI 2-sided [4.128 to 6.922] — GMR (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 3: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; GMR = 2.325, 95% CI 2-sided [1.721 to 3.140] — GMR (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 4: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; GMR = 4.221, 95% CI 2-sided [3.322 to 5.363] — GMR (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 5: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; GMR = 5.300, 95% CI 2-sided [4.243 to 6.620] — GMR (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 6: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; GMR = 1.206, 95% CI 2-sided [1.033 to 1.407] — GMR (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 7: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; GMR = 6.493, 95% CI 2-sided [4.358 to 9.674] — GMR (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-positive participants
Statistical Analysis 8: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; GMR = 5.452, 95% CI 2-sided [3.430 to 8.665] — GMR (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-positive participants
Statistical Analysis 9: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; GMR = 6.804, 95% CI 2-sided [3.928 to 11.784] — GMR (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-positive participants

7. Primary Outcome: Percentage of Participants With Seroconversion at Day 57, as Measured by PRNT50
Description: Seroconversion was defined as an increase in ZIKV-specific nAb titer from below the LLOQ to a titer equal to or above LLOQ, or an increase of at least 4-fold in ZIKV-specific nAb titer in participants with pre-existing nAb titers. LLOQ=91; ULOQ=24814.
Time Frame: Day 57
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
percentage of participants
  All Participants | 4.3 [1.74 to 8.65] | 81.0 [74.10 to 86.70] | 82.1 [75.31 to 87.67] | 39.9 [32.30 to 47.83]
  Flavivirus-seronegative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Flavivirus-seronegative Participants | 0 [0.00 to 4.74] | 86.1 [75.94 to 93.13] | 87.7 [78.47 to 93.92] | 20.4 [12.77 to 30.05]
  Flavivirus-seropositive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Flavivirus-seropositive Participants | 8.1 [3.34 to 16.05] | 75.9 [65.50 to 84.40] | 75.9 [65.02 to 84.86] | 65.7 [53.06 to 76.85]
Statistical Analysis 1: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; percentage difference = 76.69, 95% CI 2-sided [69.10 to 82.68] — Percentage Difference (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 2: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; percentage difference = 77.80, 95% CI 2-sided [70.29 to 83.67] — Percentage Difference (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 3: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; percentage difference = 35.58, 95% CI 2-sided [27.47 to 43.74] — Percentage Difference (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 4: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; percentage difference = 86.11, 95% CI 2-sided [76.25 to 92.29] — Percentage Difference (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 5: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; percentage difference = 87.65, 95% CI 2-sided [78.71 to 93.17] — Percentage Difference (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 6: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; percentage difference = 20.43, 95% CI 2-sided [13.47 to 29.75] — Percentage Difference (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 7: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; percentage difference = 67.72, 95% CI 2-sided [55.69 to 77.07] — Percentage Difference (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-positive participants
Statistical Analysis 8: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; percentage difference = 67.81, 95% CI 2-sided [55.36 to 77.44] — Percentage Difference (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-positive participants
Statistical Analysis 9: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; percentage difference = 57.53, 95% CI 2-sided [43.81 to 69.08] — Percentage Difference (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-positive participants

8. Primary Outcome: Percentage of Participants With Seroconversion at Day 57, as Measured by PRNT80
Description: as for outcome 7
Time Frame: Day 57
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
percentage of participants
  All Participants | 1.2 [0.15 to 4.36] | 76.7 [69.43 to 82.94] | 76.5 [69.25 to 82.83] | 32.5 [25.40 to 40.28]
  Flavivirus-seronegative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Flavivirus-seronegative Participants | 0 [0.00 to 4.74] | 77.8 [66.44 to 86.73] | 82.7 [72.70 to 90.22] | 9.7 [4.52 to 17.58]
  Flavivirus-seropositive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Flavivirus-seropositive Participants | 2.3 [0.28 to 8.15] | 74.7 [64.25 to 83.42] | 69.6 [58.25 to 79.47] | 65.7 [53.06 to 76.85]
Statistical Analysis 1: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; percentage difference = 75.46, 95% CI 2-sided [68.12 to 81.49] — Percentage Difference (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 2: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; percentage difference = 75.32, 95% CI 2-sided [67.94 to 81.38] — Percentage Difference (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 3: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; percentage difference = 31.29, 95% CI 2-sided [24.23 to 38.96] — Percentage Difference (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for all participants
Statistical Analysis 4: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; percentage difference = 77.78, 95% CI 2-sided [66.87 to 85.85] — Percentage Difference (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 5: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; percentage difference = 82.72, 95% CI 2-sided [73.02 to 89.43] — Percentage Difference (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 6: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; percentage difference = 9.68, 95% CI 2-sided [4.63 to 17.41] — Percentage Difference (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-negative participants
Statistical Analysis 7: Comparison: Placebo vs mRNA-1893 Low Dose (2-Dose Regimen); Test type: Other; percentage difference = 72.39, 95% CI 2-sided [61.56 to 80.83] — Percentage Difference (mRNA-1893 Low Dose [2-Dose Regimen] vs. Placebo) for flavivirus-positive participants
Statistical Analysis 8: Comparison: Placebo vs mRNA-1893 High Dose (2-Dose Regimen); Test type: Other; percentage difference = 67.29, 95% CI 2-sided [55.72 to 76.78] — Percentage Difference (mRNA-1893 High Dose [2-Dose Regimen] vs. Placebo) for flavivirus-positive participants
Statistical Analysis 9: Comparison: Placebo vs mRNA-1893 High Dose (1-Dose Regimen); Test type: Other; percentage difference = 63.35, 95% CI 2-sided [50.75 to 74.00] — Percentage Difference (mRNA-1893 High Dose [1-Dose Regimen] vs. Placebo) for flavivirus-positive participants

9. Secondary Outcome: GMT of ZIKV-Specific nAbs at Days 1, 8, 29, and 36, as Measured by PRNT50 and PRNT80
Description: as for outcome 6
Time Frame: Days 1, 8, 29, and 36
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
titer
  Day 1: All Participants by PRNT50 | 60.64 [53.33 to 68.95] | 61.21 [53.93 to 69.46] | 54.57 [49.53 to 60.13] | 59.41 [52.45 to 67.29]
  Day 8: All Participants by PRNT50: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 8: All Participants by PRNT50 | 62.15 [54.37 to 71.04] | 116.92 [90.06 to 151.81] | 105.78 [80.71 to 138.64] | 57.98 [51.17 to 65.69]
  Day 29: All Participants by PRNT50: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants by PRNT50 | 66.66 [57.15 to 77.76] | 151.34 [115.71 to 197.94] | 140.50 [107.24 to 184.08] | 59.59 [52.10 to 68.15]
  Day 36: All Participants by PRNT50: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants by PRNT50 | 58.51 [52.16 to 65.63] | 493.59 [382.88 to 636.30] | 412.24 [316.08 to 537.65] | 118.04 [89.84 to 155.09]
  Day 1: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 1: Flavivirus-negative Participants by PRNT50 | 45.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 50.76 [43.31 to 59.49] | 45.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 48.58 [44.97 to 52.48]
  Day 8: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants by PRNT50 | 45.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 50.24 [43.73 to 57.71] | 48.05 [44.03 to 52.43] | 50.30 [45.07 to 56.15]
  Day 29: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants by PRNT50 | 46.45 [44.58 to 48.39] | 57.81 [48.16 to 69.40] | 67.45 [56.47 to 80.56] | 48.85 [45.24 to 52.75]
  Day 36: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants by PRNT50 | 45.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 478.42 [346.32 to 660.91] | 344.02 [249.51 to 474.33] | 56.46 [46.29 to 68.86]
  Day 1: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 1: Flavivirus-positive Participants by PRNT50 | 78.42 [62.17 to 98.91] | 72.45 [59.72 to 87.88] | 66.06 [54.52 to 80.03] | 79.50 [60.53 to 104.40]
  Day 8: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT50 | 81.87 [64.46 to 103.98] | 245.67 [161.42 to 373.91] | 245.31 [150.29 to 400.42] | 71.60 [55.17 to 92.92]
  Day 29: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants by PRNT50 | 92.15 [70.05 to 121.22] | 350.77 [234.46 to 524.78] | 295.81 [184.73 to 473.71] | 79.46 [58.87 to 107.25]
  Day 36: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT50 | 73.48 [59.61 to 90.57] | 507.03 [340.84 to 754.26] | 487.78 [315.43 to 754.30] | 339.16 [203.88 to 564.20]
  Day 1: All Participants by PRNT80 | 21.06 [18.82 to 23.58] | 21.23 [19.13 to 23.56] | 18.94 [17.56 to 20.42] | 19.60 [17.84 to 21.54]
  Day 8: All Participants by PRNT80: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 8: All Participants by PRNT80 | 20.50 [18.46 to 22.77] | 40.88 [31.55 to 52.97] | 37.44 [28.52 to 49.16] | 20.10 [18.01 to 22.42]
  Day 29: All Participants by PRNT80: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants by PRNT80 | 21.07 [18.94 to 23.44] | 49.95 [38.14 to 65.42] | 43.46 [33.06 to 57.13] | 19.72 [17.83 to 21.82]
  Day 36: All Participants by PRNT80: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants by PRNT80 | 20.40 [18.42 to 22.59] | 124.30 [97.25 to 158.87] | 121.27 [93.24 to 157.71] | 39.69 [30.34 to 51.92]
  Day 1: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 1: Flavivirus-negative Participants by PRNT80 | 16.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 18.06 [15.91 to 20.49] | 16.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 17.63 [16.28 to 19.10]
  Day 8: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants by PRNT80 | 16.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 18.43 [15.78 to 21.52] | 17.24 [15.80 to 18.81] | 17.58 [16.22 to 19.05]
  Day 29: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants by PRNT80 | 16.95 [16.07 to 17.88] | 18.75 [16.15 to 21.75] | 19.06 [16.73 to 21.72] | 17.64 [16.25 to 19.15]
  Day 36: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants by PRNT80 | 16.50 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 95.88 [71.94 to 127.78] | 89.62 [66.16 to 121.40] | 19.02 [16.09 to 22.48]
  Day 1: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 1: Flavivirus-positive Participants by PRNT80 | 26.21 [21.36 to 32.16] | 24.56 [20.91 to 28.85] | 21.89 [18.84 to 25.42] | 22.89 [18.78 to 27.89]
  Day 8: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT80 | 24.84 [20.54 to 30.04] | 82.41 [54.22 to 125.26] | 85.57 [52.06 to 140.65] | 24.49 [19.27 to 31.12]
  Day 29: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants by PRNT80 | 25.61 [21.21 to 30.93] | 116.95 [77.36 to 176.79] | 99.92 [61.83 to 161.47] | 23.21 [18.71 to 28.79]
  Day 36: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT80 | 24.73 [20.52 to 29.81] | 156.24 [105.60 to 231.16] | 161.96 [104.84 to 250.22] | 113.38 [67.59 to 190.20]

10. Secondary Outcome: GMT of ZIKV-Specific nAbs at Days 1, 8, 29, 36, and 57, as Measured by Microneutralization (MN)
Description: Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values that were greater than the ULOQ were converted to the ULOQ. LLOQ=28; ULOQ=11589. 95% CI was calculated based on the t-distribution of the log-transformed values, then back transformed to the original scale for presentation.
Time Frame: Days 1, 8, 29, 36, and 57
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
titer
  Day 1: All Participants | 30.54 [24.08 to 38.73] | 32.98 [26.18 to 41.55] | 25.31 [20.43 to 31.36] | 27.94 [22.45 to 34.78]
  Day 8: All Participants: number analyzed (Participants) | 162 | 163 | 162 | 163
  Day 8: All Participants | 27.99 [22.52 to 34.80] | 76.17 [52.37 to 110.79] | 80.70 [55.40 to 117.55] | 24.68 [20.43 to 29.80]
  Day 29: All Participants: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants | 32.05 [25.20 to 40.75] | 489.20 [365.80 to 654.24] | 544.38 [416.59 to 711.36] | 28.61 [22.85 to 35.83]
  Day 36: All Participants: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants | 27.74 [22.42 to 34.32] | 1318.97 [1068.49 to 1628.15] | 1380.12 [1109.40 to 1716.91] | 81.79 [56.62 to 118.15]
  Day 57: All Participants | 31.60 [24.81 to 40.24] | 2261.02 [1903.39 to 2685.84] | 2270.12 [1907.12 to 2702.22] | 643.02 [491.83 to 840.67]
  Day 1: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 1: Flavivirus-negative Participants | 14.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 16.25 [13.69 to 19.30] | 14.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 15.99 [13.66 to 18.72]
  Day 8: Flavivirus-negative Participants: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants | 14.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 17.73 [13.79 to 22.80] | 20.22 [16.32 to 25.04] | 15.66 [13.76 to 17.82]
  Day 29: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants | 14.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 200.15 [148.92 to 268.99] | 285.93 [211.77 to 386.07] | 16.92 [13.99 to 20.47]
  Day 36: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants | 14.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 1428.20 [1110.81 to 1836.29] | 1237.86 [923.46 to 1659.31] | 23.16 [17.78 to 30.17]
  Day 57: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 57: Flavivirus-negative Participants | 14.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 2291.24 [1821.46 to 2882.20] | 2235.55 [1826.02 to 2736.92] | 280.91 [211.58 to 372.97]
  Day 1: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 1: Flavivirus-positive Participants | 61.39 [41.21 to 91.45] | 61.63 [42.84 to 88.66] | 47.15 [31.65 to 70.26] | 62.55 [41.06 to 95.28]
  Day 8: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 8: Flavivirus-positive Participants | 51.65 [35.80 to 74.50] | 275.14 [159.62 to 474.24] | 348.73 [193.37 to 628.91] | 47.58 [32.70 to 69.24]
  Day 29: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants | 67.27 [45.25 to 99.98] | 1040.81 [680.49 to 1591.92] | 1067.67 [711.80 to 1601.47] | 61.27 [40.18 to 93.42]
  Day 36: Flavivirus-positive Participants: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants | 51.54 [35.96 to 73.87] | 1260.49 [898.36 to 1768.61] | 1504.49 [1076.56 to 2102.53] | 493.88 [273.73 to 891.11]
  Day 57: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 57: Flavivirus-positive Participants | 65.50 [43.82 to 97.91] | 2246.56 [1727.41 to 2921.74] | 2253.47 [1681.38 to 3020.20] | 2002.83 [1367.92 to 2932.43]

11. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of ZIKV-Specific nAbs at Days 8, 29, 36, and 57, as Measured by PRNT50 and PRNT80
Description: Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values that were greater than the ULOQ were converted to the ULOQ. LLOQ=91; ULOQ=248. 95% CI was calculated based on the t-distribution of the difference in the log-transformed values, then back transformed to the original scale for presentation.
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
ratio
  Day 8: All Participants by PRNT50: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 8: All Participants by PRNT50 | 1.02 [0.94 to 1.11] | 1.91 [1.55 to 2.36] | 1.94 [1.54 to 2.43] | 0.98 [0.87 to 1.1]
  Day 29: All Participants by PRNT50: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants by PRNT50 | 1.10 [0.99 to 1.22] | 2.47 [1.98 to 3.08] | 2.57 [2.05 to 3.23] | 1.00 [0.93 to 1.08]
  Day 36: All Participants by PRNT50: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants by PRNT50 | 0.96 [0.89 to 1.04] | 8.06 [6.30 to 10.32] | 7.55 [5.91 to 9.63] | 1.98 [1.59 to 2.48]
  Day 57: All Participants by PRNT50 | 1.01 [0.93 to 1.09] | 6.98 [5.68 to 8.59] | 7.97 [6.45 to 9.85] | 2.75 [2.18 to 3.46]
  Day 8: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants by PRNT50 | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 0.99 [0.95 to 1.03] | 1.06 [0.97 to 1.15] | 1.04 [0.95 to 1.13]
  Day 29: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants by PRNT50 | 1.02 [0.98 to 1.06] | 1.14 [1.02 to 1.27] | 1.48 [1.24 to 1.77] | 1.01 [0.98 to 1.03]
  Day 36: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants by PRNT50 | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 9.43 [6.70 to 13.26] | 7.56 [5.48 to 10.42] | 1.16 [1.00 to 1.34]
  Day 57: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 57: Flavivirus-negative Participants by PRNT50 | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 6.46 [4.92 to 8.48] | 7.98 [6.11 to 10.43] | 1.42 [1.20 to 1.68]
  Day 8: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT50 | 1.04 [0.90 to 1.21] | 3.39 [2.37 to 4.84] | 3.70 [2.44 to 5.61] | 0.90 [0.69 to 1.19]
  Day 29: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants by PRNT50 | 1.18 [0.96 to 1.43] | 4.84 [3.42 to 6.85] | 4.48 [3.03 to 6.61] | 1.00 [0.83 to 1.20]
  Day 36: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT50 | 0.93 [0.81 to 1.08] | 7.00 [4.85 to 10.09] | 7.38 [5.04 to 10.81] | 4.27 [2.74 to 6.64]
  Day 57: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 57: Flavivirus-positive Participants by PRNT50 | 1.01 [0.87 to 1.19] | 7.44 [5.40 to 10.25] | 7.60 [5.42 to 10.66] | 7.03 [4.61 to 10.70]
  Day 8: All Participants by PRNT80: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 8: All Participants by PRNT80 | 0.97 [0.94 to 1.01] | 1.93 [1.57 to 2.36] | 1.98 [1.57 to 2.49] | 1.03 [0.98 to 1.09]
  Day 29: All Participants by PRNT80: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants by PRNT80 | 1.00 [0.96 to 1.04] | 2.35 [1.88 to 2.94] | 2.29 [1.82 to 2.90] | 1.01 [0.99 to 1.03]
  Day 36: All Participants by PRNT80: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants by PRNT80 | 0.97 [0.92 to 1.01] | 5.85 [4.72 to 7.27] | 6.40 [5.06 to 8.09] | 2.02 [1.63 to 2.52]
  Day 57: All Participants by PRNT80 | 0.99 [0.94 to 1.04] | 5.21 [4.28 to 6.33] | 5.87 [4.79 to 7.21] | 2.47 [1.94 to 3.13]
  Day 8: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants by PRNT80 | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 1.02 [0.99 to 1.05] | 1.04 [0.96 to 1.14] | 1.00 [0.98 to 1.01]
  Day 29: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants by PRNT80 | 1.03 [0.97 to 1.08] | 1.04 [0.97 to 1.11] | 1.16 [1.01 to 1.32] | 1.00 [0.99 to 1.01]
  Day 36: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants by PRNT80 | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 5.31 [4.02 to 7.02] | 5.43 [4.01 to 7.36] | 1.08 [0.99 to 1.18]
  Day 57: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 57: Flavivirus-negative Participants by PRNT80 | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 3.86 [3.03 to 4.91] | 5.30 [4.24 to 6.62] | 1.13 [1.04 to 1.23]
  Day 8: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT80 | 0.95 [0.89 to 1.01] | 3.36 [2.38 to 4.74] | 3.90 [2.55 to 5.94] | 1.09 [0.95 to 1.24]
  Day 29: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants by PRNT80 | 0.98 [0.93 to 1.03] | 4.76 [3.34 to 6.79] | 4.57 [3.05 to 6.84] | 1.01 [0.96 to 1.07]
  Day 36: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT80 | 0.94 [0.86 to 1.03] | 6.36 [4.55 to 8.90] | 7.40 [5.12 to 10.69] | 4.95 [3.21 to 7.65]
  Day 57: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 57: Flavivirus-positive Participants by PRNT80 | 0.98 [0.89 to 1.07] | 6.77 [5.01 to 9.15] | 6.38 [4.48 to 9.08] | 7.61 [4.84 to 11.96]

12. Secondary Outcome: GMFR of ZIKV-Specific nAbs at Days 8, 29, 36, and 57, as Measured by MN
Description: Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values that were greater than the ULOQ were converted to the ULOQ. LLOQ=28; ULOQ=11589. 95% CI was calculated based on the t-distribution of the difference in the log-transformed values, then back transformed to the original scale for presentation.
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
ratio
  Day 8: All Participants: number analyzed (Participants) | 162 | 163 | 162 | 163
  Day 8: All Participants | 0.91 [0.85 to 0.97] | 2.31 [1.87 to 2.85] | 3.19 [2.50 to 4.06] | 0.88 [0.82 to 0.95]
  Day 29: All Participants: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants | 1.05 [0.97 to 1.13] | 14.75 [12.03 to 18.09] | 21.51 [17.65 to 26.21] | 1.02 [0.96 to 1.09]
  Day 36: All Participants: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants | 0.90 [0.84 to 0.97] | 39.99 [31.83 to 50.25] | 54.33 [43.90 to 67.23] | 2.91 [2.34 to 3.64]
  Day 57: All Participants | 1.03 [0.96 to 1.12] | 68.55 [54.98 to 85.48] | 89.69 [72.82 to 110.47] | 23.01 [18.89 to 28.03]
  Day 8: Flavivirus-negative Participants: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 1.09 [0.95 to 1.25] | 1.44 [1.17 to 1.79] | 0.98 [0.94 to 1.02]
  Day 29: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 12.29 [9.46 to 15.97] | 20.42 [15.13 to 27.58] | 1.06 [0.96 to 1.16]
  Day 36: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 87.88 [67.32 to 114.73] | 88.42 [65.96 to 118.52] | 1.45 [1.22 to 1.72]
  Day 57: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 57: Flavivirus-negative Participants | 1.00 [NA to NA] — Due to not enough variability in the values, the CI (upper and lower limit) could not be calculated. | 140.99 [108.71 to 182.85] | 159.68 [130.43 to 195.49] | 17.57 [13.53 to 22.80]
  Day 8: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 8: Flavivirus-positive Participants | 0.84 [0.75 to 0.95] | 4.46 [3.24 to 6.15] | 7.40 [5.12 to 10.68] | 0.76 [0.65 to 0.90]
  Day 29: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants | 1.10 [0.94 to 1.27] | 16.89 [12.39 to 23.02] | 22.64 [17.39 to 29.48] | 0.98 [0.89 to 1.07]
  Day 36: Flavivirus-positive Participants: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants | 0.83 [0.73 to 0.94] | 20.45 [15.07 to 27.76] | 31.91 [24.26 to 41.95] | 7.90 [5.45 to 11.43]
  Day 57: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 57: Flavivirus-positive Participants | 1.07 [0.92 to 1.24] | 36.45 [27.11 to 49.02] | 47.79 [34.69 to 65.84] | 32.02 [23.77 to 43.13]

13. Secondary Outcome: Percentage of Participants With Seroconversion at Days 8, 29, and 36, as Measured by PRNT50 and PRNT80
Description: as for outcome 7
Time Frame: Days 8, 29, and 36
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
percentage of participants
  Day 8: All Participants by PRNT50: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 8: All Participants by PRNT50 | 3.1 [1.01 to 7.06] | 20.9 [14.90 to 27.91] | 21.1 [15.09 to 28.24] | 4.3 [1.75 to 8.70]
  Day 29: All Participants by PRNT50: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants by PRNT50 | 6.7 [3.42 to 11.75] | 33.3 [26.13 to 41.16] | 38.3 [30.76 to 46.22] | 3.7 [1.36 to 7.84]
  Day 36: All Participants by PRNT50: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants by PRNT50 | 1.9 [0.38 to 5.32] | 76.1 [68.78 to 82.40] | 75.2 [67.74 to 81.62] | 21.0 [14.99 to 28.07]
  Day 8: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants by PRNT50 | 0 [0.00 to 4.80] | 0 [0.00 to 4.99] | 2.5 [0.30 to 8.64] | 1.1 [0.03 to 5.85]
  Day 29: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants by PRNT50 | 1.3 [0.03 to 7.11] | 8.5 [3.16 to 17.49] | 25.9 [16.82 to 36.86] | 1.1 [0.03 to 5.85]
  Day 36: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants by PRNT50 | 0 [0.00 to 4.74] | 86.1 [75.94 to 93.13] | 78.8 [68.17 to 87.11] | 4.3 [1.20 to 10.76]
  Day 8: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT50 | 5.8 [1.91 to 13.05] | 39.1 [28.79 to 50.13] | 41.0 [30.01 to 52.75] | 9.1 [3.41 to 18.74]
  Day 29: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants by PRNT50 | 11.6 [5.72 to 20.35] | 55.2 [44.13 to 65.85] | 50.6 [39.14 to 62.08] | 7.5 [2.47 to 16.56]
  Day 36: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT50 | 3.5 [0.73 to 9.97] | 66.7 [55.75 to 76.42] | 70.9 [59.58 to 80.57] | 44.8 [32.60 to 57.42]
  Day 8: All Participants by PRNT80: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 8: All Participants by PRNT80 | 0 [0.00 to 2.25] | 19.6 [13.83 to 26.57] | 19.3 [13.47 to 26.20] | 1.2 [0.15 to 4.39]
  Day 29: All Participants by PRNT80: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants by PRNT80 | 1.2 [0.15 to 4.36] | 31.5 [24.42 to 39.23] | 29.0 [22.16 to 36.65] | 0 [0.00 to 2.24]
  Day 36: All Participants by PRNT80: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants by PRNT80 | 1.2 [0.15 to 4.39] | 72.4 [64.86 to 79.10] | 72.0 [64.44 to 78.83] | 22.8 [16.62 to 30.08]
  Day 8: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants by PRNT80 | 0 [0.00 to 4.80] | 0 [0.00 to 4.99] | 1.2 [0.03 to 6.69] | 0 [0.00 to 3.89]
  Day 29: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants by PRNT80 | 1.3 [0.03 to 7.11] | 2.8 [0.34 to 9.81] | 7.4 [2.77 to 15.43] | 0 [0.00 to 3.89]
  Day 36: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants by PRNT80 | 0 [0.00 to 4.74] | 75.0 [63.40 to 84.46] | 71.3 [60.05 to 80.82] | 3.3 [0.68 to 9.23]
  Day 8: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT80 | 0 [0.00 to 4.20] | 36.8 [26.69 to 47.80] | 38.5 [27.66 to 50.17] | 3.0 [0.37 to 10.52]
  Day 29: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants by PRNT80 | 1.2 [0.03 to 6.31] | 56.3 [45.26 to 66.94] | 50.6 [39.14 to 62.08] | 0 [0.00 to 5.36]
  Day 36: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT80 | 2.4 [0.29 to 8.24] | 69.0 [58.14 to 78.45] | 72.2 [60.93 to 81.65] | 50.7 [38.24 to 63.18]

14. Secondary Outcome: Percentage of Participants With Seroconversion at Days 8, 29, 36, and 57, as Measured by MN
Description: Seroconversion was defined as an increase in ZIKV-specific nAb titer from below the LLOQ to a titer equal to or above LLOQ, or an increase of at least 4-fold in ZIKV-specific nAb titer in participants with pre-existing nAb titers. LLOQ=28; ULOQ=11589.
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 163 | 163 | 162 | 163
percentage of participants
  Day 8: All Participants: number analyzed (Participants) | 162 | 163 | 162 | 163
  Day 8: All Participants | 1.2 [0.15 to 4.39] | 35.0 [27.68 to 42.82] | 41.4 [33.69 to 49.35] | 1.2 [0.15 to 4.36]
  Day 29: All Participants: number analyzed (Participants) | 163 | 162 | 162 | 163
  Day 29: All Participants | 1.8 [0.38 to 5.28] | 93.2 [88.18 to 96.56] | 95.7 [91.30 to 98.25] | 1.8 [0.38 to 5.28]
  Day 36: All Participants: number analyzed (Participants) | 162 | 163 | 161 | 162
  Day 36: All Participants | 1.2 [0.15 to 4.39] | 92.6 [87.49 to 96.14] | 96.3 [92.07 to 98.62] | 40.7 [33.10 to 48.73]
  Day 57: All Participants | 1.8 [0.38 to 5.28] | 95.7 [91.35 to 98.26] | 97.5 [93.80 to 99.32] | 95.7 [91.35 to 98.26]
  Day 8: Flavivirus-negative Participants: number analyzed (Participants) | 75 | 72 | 81 | 93
  Day 8: Flavivirus-negative Participants | 0 [0.00 to 4.80] | 8.3 [3.12 to 17.26] | 16.0 [8.83 to 25.88] | 0 [0.00 to 3.89]
  Day 29: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 71 | 81 | 93
  Day 29: Flavivirus-negative Participants | 0 [0.00 to 4.74] | 97.2 [90.19 to 99.66] | 95.1 [87.84 to 98.64] | 1.1 [0.03 to 5.85]
  Day 36: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 72 | 80 | 92
  Day 36: Flavivirus-negative Participants | 0 [0.00 to 4.74] | 98.6 [92.50 to 99.96] | 97.5 [91.26 to 99.70] | 18.5 [11.15 to 27.93]
  Day 57: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 72 | 81 | 93
  Day 57: Flavivirus-negative Participants | 0 [0.00 to 4.74] | 98.6 [92.50 to 99.96] | 100.0 [95.55 to 100.0] | 94.6 [87.90 to 98.23]
  Day 8: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 8: Flavivirus-positive Participants | 2.3 [0.28 to 8.15] | 58.6 [47.55 to 69.08] | 68.4 [56.92 to 78.37] | 3.0 [0.36 to 10.37]
  Day 29: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 29: Flavivirus-positive Participants | 3.5 [0.73 to 9.86] | 89.7 [81.27 to 95.16] | 96.2 [89.30 to 99.21] | 3.0 [0.36 to 10.37]
  Day 36: Flavivirus-positive Participants: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants | 2.4 [0.29 to 8.24] | 87.4 [78.50 to 93.52] | 94.9 [87.54 to 98.60] | 71.6 [59.31 to 81.99]
  Day 57: Flavivirus-positive Participants: number analyzed (Participants) | 86 | 87 | 79 | 67
  Day 57: Flavivirus-positive Participants | 3.5 [0.73 to 9.86] | 93.1 [85.59 to 97.43] | 94.9 [87.54 to 98.60] | 97.0 [89.63 to 99.64]

15. Secondary Outcome: Percentage of Initially Seronegative Participants With a Seroresponse at Days 8, 29, and 36, as Measured by PRNT50 and PRNT80
Description: Seroresponse was defined as an increase in ZIKV-specific nAb titer from below the LLOQ to greater than or equal to the LLOQ. LLOQ=91; ULOQ=24814.
Time Frame: Days 8, 29, and 36
Population: The PPAMI included all participants who received any study injection, who did not have major protocol deviations that impacted AMI response, and who complied with the injection schedule and timing of immunogenicity blood sampling to have post-injection results available for at least 1 assay component of AMI at the corresponding visit. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified categories.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 76 | 70 | 81 | 93
percentage of participants
  Day 8: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 75 | 70 | 81 | 93
  Day 8: Flavivirus-negative Participants by PRNT50 | 0 [0.00 to 4.80] | 0 [0.00 to 5.13] | 2.5 [0.30 to 8.64] | 1.1 [0.03 to 6.04]
  Day 29: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 69 | 81 | 93
  Day 29: Flavivirus-negative Participants by PRNT50 | 1.3 [0.03 to 7.11] | 8.7 [3.26 to 17.97] | 25.9 [16.82 to 36.86] | 1.1 [0.03 to 6.04]
  Day 36: Flavivirus-negative Participants by PRNT50: number analyzed (Participants) | 76 | 70 | 80 | 89
  Day 36: Flavivirus-negative Participants by PRNT50 | 0 [0.00 to 4.74] | 88.6 [78.72 to 94.93] | 78.8 [68.17 to 87.11] | 2.2 [0.27 to 7.88]
  Day 8: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 75 | 70 | 81 | 90
  Day 8: Flavivirus-negative Participants by PRNT80 | 0 [0.00 to 4.80] | 0 [0.00 to 5.13] | 1.2 [0.03 to 6.69] | 0 [0.00 to 4.02]
  Day 29: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 69 | 81 | 90
  Day 29: Flavivirus-negative Participants by PRNT80 | 1.3 [0.03 to 7.11] | 2.9 [0.35 to 10.08] | 7.4 [2.77 to 15.43] | 0 [0.00 to 4.02]
  Day 36: Flavivirus-negative Participants by PRNT80: number analyzed (Participants) | 76 | 70 | 80 | 89
  Day 36: Flavivirus-negative Participants by PRNT80 | 0 [0.00 to 4.74] | 77.1 [65.55 to 86.33] | 71.3 [60.05 to 80.82] | 0 [0.00 to 4.06]

16. Secondary Outcome: Percentage of Initially Seronegative Participants With a Seroresponse at Days 8, 29, 36, and 57, as Measured by MN
Description: Seroresponse was defined as an increase in ZIKV-specific nAb titer from below the LLOQ to greater than or equal to the LLOQ. LLOQ=28; ULOQ=11589.
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 76 | 69 | 81 | 90
percentage of participants
  Day 8: Flavivirus-negative Participants: number analyzed (Participants) | 75 | 69 | 81 | 90
  Day 8: Flavivirus-negative Participants | 0 [0.00 to 4.80] | 5.8 [1.60 to 14.18] | 16.0 [8.83 to 25.88] | 0 [0.00 to 4.02]
  Day 29: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 68 | 81 | 90
  Day 29: Flavivirus-negative Participants | 0 [0.00 to 4.74] | 97.1 [89.78 to 99.64] | 95.1 [87.84 to 98.64] | 1.1 [0.03 to 6.04]
  Day 36: Flavivirus-negative Participants: number analyzed (Participants) | 76 | 69 | 80 | 89
  Day 36: Flavivirus-negative Participants | 0 [0.00 to 4.74] | 98.6 [92.19 to 99.96] | 97.5 [91.26 to 99.70] | 15.7 [8.88 to 24.98]
  Day 57: Flavivirus-negative Participants | 0 [0.00 to 4.74] | 98.6 [92.19 to 99.96] | 100.0 [95.55 to 100.0] | 94.4 [87.51 to 98.17]

17. Secondary Outcome: Percentage of Initially Seropositive Participants With a 2-Fold Increase in ZIKV-Specific nAb Titers as Compared With Baseline, as Measured by PRNT50 and PRNT80
Description: ≥2-fold increase from baseline was defined as a ≥2 * LLOQ for participants with baseline undetectable antibody titer, or a 2-times or higher ratio in participants with pre-existing nAb titers. LLOQ=91
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 86 | 87 | 79 | 67
percentage of participants
  Day 8: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT50 | 8.1 [3.34 to 16.05] | 41.4 [30.92 to 52.45] | 38.5 [27.66 to 50.17] | 6.1 [1.68 to 14.80]
  Day 29: Flavivirus-positive Participants by PRNT50 | 10.5 [4.90 to 18.94] | 55.2 [44.13 to 65.85] | 44.3 [33.12 to 55.92] | 6.0 [1.65 to 14.59]
  Day 36: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT50 | 4.7 [1.30 to 11.61] | 60.9 [49.87 to 71.21] | 63.3 [51.69 to 73.86] | 46.3 [34.00 to 58.88]
  Day 57: Flavivirus-positive Participants by PRNT50 | 5.8 [1.91 to 13.05] | 63.2 [52.20 to 73.31] | 63.3 [51.69 to 73.86] | 62.7 [50.01 to 74.20]
  Day 8: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT80 | 0 [0.00 to 4.20] | 40.2 [29.85 to 51.29] | 38.5 [27.66 to 50.17] | 4.5 [0.95 to 12.71]
  Day 29: Flavivirus-positive Participants by PRNT80 | 0 [0.00 to 4.20] | 49.4 [38.53 to 60.36] | 43.0 [31.94 to 54.67] | 1.5 [0.04 to 8.04]
  Day 36: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT80 | 1.2 [0.03 to 6.38] | 63.2 [52.20 to 73.31] | 62.0 [50.41 to 72.72] | 50.7 [38.24 to 63.18]
  Day 57: Flavivirus-positive Participants by PRNT80 | 3.5 [0.73 to 9.86] | 63.2 [52.20 to 73.31] | 60.8 [49.13 to 71.56] | 61.2 [48.50 to 72.86]

18. Secondary Outcome: Percentage of Initially Seropositive Participants With a 4-Fold Increase in ZIKV-Specific nAb Titers as Compared With Baseline, as Measured by PRNT50 and PRNT80
Description: ≥4-fold increase from baseline was defined as a ≥4 * LLOQ for participants with baseline undetectable antibody titer, or a 4-times or higher ratio in participants with pre-existing nAb titers. LLOQ=91
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 86 | 87 | 79 | 67
percentage of participants
  Day 8: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT50 | 2.3 [0.28 to 8.15] | 35.6 [25.65 to 46.62] | 35.9 [25.34 to 47.56] | 4.5 [0.95 to 12.71]
  Day 29: Flavivirus-positive Participants by PRNT50 | 7.0 [2.60 to 14.57] | 42.5 [31.99 to 53.59] | 40.5 [29.60 to 52.15] | 4.5 [0.93 to 12.53]
  Day 36: Flavivirus-positive Participants by PRNT50: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT50 | 1.2 [0.03 to 6.38] | 50.6 [39.64 to 61.47] | 50.6 [39.14 to 62.08] | 38.8 [27.14 to 51.50]
  Day 57: Flavivirus-positive Participants by PRNT50 | 2.3 [0.28 to 8.15] | 52.9 [41.87 to 63.67] | 48.1 [36.71 to 59.64] | 47.8 [35.40 to 60.33]
  Day 8: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 86 | 87 | 78 | 66
  Day 8: Flavivirus-positive Participants by PRNT80 | 0 [0.00 to 4.20] | 35.6 [25.65 to 46.62] | 33.3 [23.06 to 44.92] | 1.5 [0.04 to 8.16]
  Day 29: Flavivirus-positive Participants by PRNT80 | 0 [0.00 to 4.20] | 40.2 [29.85 to 51.29] | 38.0 [27.28 to 49.59] | 0 [0.00 to 5.36]
  Day 36: Flavivirus-positive Participants by PRNT80: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants by PRNT80 | 0 [0.00 to 4.25] | 50.6 [39.64 to 61.47] | 50.6 [39.14 to 62.08] | 43.3 [31.22 to 55.96]
  Day 57: Flavivirus-positive Participants by PRNT80 | 1.2 [0.03 to 6.31] | 50.6 [39.64 to 61.47] | 43.0 [31.94 to 54.67] | 49.3 [36.82 to 61.76]

19. Secondary Outcome: Percentage of Initially Seropositive Participants With a 2-Fold Increase in ZIKV-Specific nAb Titers as Compared With Baseline, as Measured by MN
Description: ≥2-fold increase from baseline was defined as a ≥2 * LLOQ for participants with baseline undetectable antibody titer, or a 2-times or higher ratio in participants with pre-existing nAb titers. LLOQ=28.
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 86 | 87 | 79 | 67
percentage of participants
  Day 8: Flavivirus-positive Participants | 3.5 [0.73 to 9.86] | 58.6 [47.55 to 69.08] | 63.3 [51.69 to 73.86] | 4.5 [0.93 to 12.53]
  Day 29: Flavivirus-positive Participants | 2.3 [0.28 to 8.15] | 87.4 [78.50 to 93.52] | 96.2 [89.30 to 99.21] | 0 [0.00 to 5.36]
  Day 36: Flavivirus-positive Participants: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants | 4.7 [1.30 to 11.61] | 92.0 [84.12 to 96.70] | 97.5 [91.15 to 99.69] | 71.6 [59.31 to 81.99]
  Day 57: Flavivirus-positive Participants | 2.3 [0.28 to 8.15] | 97.7 [91.94 to 99.72] | 98.7 [93.15 to 99.97] | 100.0 [94.64 to 100.00]

20. Secondary Outcome: Percentage of Initially Seropositive Participants With a 4-Fold Increase in ZIKV-Specific nAb Titers as Compared With Baseline, as Measured by MN
Description: ≥4-fold increase from baseline was defined as a ≥4 * LLOQ for participants with baseline undetectable antibody titer, or a 4-times or higher ratio in participants with pre-existing nAb titers. LLOQ=28.
Time Frame: Days 8, 29, 36, and 57
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | mRNA-1893 Low Dose (2-Dose Regimen) | mRNA-1893 High Dose (2-Dose Regimen) | mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 86 | 87 | 79 | 67
percentage of participants
  Day 8: Flavivirus-positive Participants | 2.3 [0.28 to 8.15] | 43.7 [33.06 to 54.74] | 50.6 [39.14 to 62.08] | 1.5 [0.04 to 8.04]
  Day 29: Flavivirus-positive Participants | 2.3 [0.28 to 8.15] | 79.3 [69.29 to 87.25] | 87.3 [77.95 to 93.76] | 0 [0.00 to 5.36]
  Day 36: Flavivirus-positive Participants: number analyzed (Participants) | 85 | 87 | 79 | 67
  Day 36: Flavivirus-positive Participants | 1.2 [0.03 to 6.38] | 81.6 [71.86 to 89.11] | 92.4 [84.20 to 97.16] | 58.2 [45.52 to 70.15]
  Day 57: Flavivirus-positive Participants | 2.3 [0.28 to 8.15] | 93.1 [85.59 to 97.43] | 93.7 [85.84 to 97.91] | 92.5 [83.44 to 97.53]

21. Other Pre Specified Outcome: Number of Deaths Related to Study Drug
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, irrespective of its perceived relationship to the study drug. The Investigator assessed the causality by determining whether there was a reasonable possibility that the death was related to the study drug, using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable AND/OR the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable.
Time Frame: Day 1 through Day 196 for Main Study and Day 197 through Day 700 for Extension Period
Population: The Randomized Set included all participants who were randomized in the study, regardless of the participant's treatment status in the study. One participant who was randomized at two sites and received two injections was kept in both arms (Randomized to mRNA-1893 High Dose [2-Dose Regimen] and mRNA-1893 Low Dose [2-Dose Regimen]) in Randomized Set for collection and reporting data.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Placebo | Main Study: mRNA-1893 Low Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (1-Dose Regimen) | Extension Period: Placebo | Extension Period: mRNA-1893 Low Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (1-Dose Regimen)
Number analyzed (Participants) | 203 | 202 | 203 | 201 | 113 | 109 | 104 | 116
Participants
  Deaths | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Deaths Related to Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were collected from Day 1 through Day 196 for Main Study and Day 197 through Day 700 for Extension Period. Other (not including serious) unsolicited adverse events were collected up to 28 days after study injection (that is, Day 1 up to Day 57) unless they met the criteria for AESIs, MAAEs or AEs led to discontinuation.
Description: The all-cause mortality was based on the randomized set. The serious and other (not including serious) adverse events were based on the safety set which consisted of all randomized participants who received any study injection. One participant who was randomized at two sites and received two injections was kept in both arms (Randomized to mRNA-1893 High Dose [2-Dose Regimen] and mRNA-1893 Low Dose [2-Dose Regimen]) in Randomized Set and Safety Set for collection and reporting data.
Arm/Group | Main Study: Placebo | Main Study: mRNA-1893 Low Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (2-Dose Regimen) | Main Study: mRNA-1893 High Dose (1-Dose Regimen) | Extension Period: Placebo | Extension Period: mRNA-1893 Low Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (2-Dose Regimen) | Extension Period: mRNA-1893 High Dose (1-Dose Regimen)
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/202 | 0/203 | 1/201 | 0/113 | 1/109 | 0/104 | 0/116
Serious Adverse Events (participants affected / at risk) | 5/201 | 2/202 | 4/202 | 7/198 | 5/113 | 4/109 | 5/104 | 7/116
Other Adverse Events (participants affected / at risk) | 18/201 | 20/202 | 24/202 | 16/198 | 8/113 | 5/109 | 8/104 | 10/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Placebo (N=201) | Main Study: mRNA-1893 Low Dose (2-Dose Regimen) (N=202) | Main Study: mRNA-1893 High Dose (2-Dose Regimen) (N=202) | Main Study: mRNA-1893 High Dose (1-Dose Regimen) (N=198) | Extension Period: Placebo (N=113) | Extension Period: mRNA-1893 Low Dose (2-Dose Regimen) (N=109) | Extension Period: mRNA-1893 High Dose (2-Dose Regimen) (N=104) | Extension Period: mRNA-1893 High Dose (1-Dose Regimen) (N=116)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Factitious disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff tear arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRCA1 gene mutation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Placebo (N=201) | Main Study: mRNA-1893 Low Dose (2-Dose Regimen) (N=202) | Main Study: mRNA-1893 High Dose (2-Dose Regimen) (N=202) | Main Study: mRNA-1893 High Dose (1-Dose Regimen) (N=198) | Extension Period: Placebo (N=113) | Extension Period: mRNA-1893 Low Dose (2-Dose Regimen) (N=109) | Extension Period: mRNA-1893 High Dose (2-Dose Regimen) (N=104) | Extension Period: mRNA-1893 High Dose (1-Dose Regimen) (N=116)
COVID-19 (Infections and infestations) | 12 (12) | 13 (13) | 22 (23) | 12 (12) | 3 (3) | 0 (0) | 3 (3) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 8 (8) | 2 (2) | 5 (6) | 6 (6) | 5 (5) | 5 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT04917861/Prot_001.pdf
  • Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT04917861/SAP_002.pdf
  • Informed Consent Form (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04917861/ICF_000.pdf